CLINICAL TRIAL: NCT02383628
Title: Endoscopic Perfusion Utilizing ICG Fluorescence Technology
Acronym: ICG
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Paul Gardner, Associate Professor, University of Pittsburgh
Other Study IDs: PRO13110107
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Quality of Life
Keywords: ICG Dye; endoscopic neurosurgery; tissue perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the study is to evaluate the efficacy of indocyanine green (ICG) endoscopy to evaluate tissue perfusion during endoscopic neurosurgery. This includes patients with pituitary and intracranial tumors and treatment of vascular abnormalities such as aneurysms and compressive syndromes. ICG will be evaluated to determine the value of the additional visual information supplied during the treatment of these pathologies.

DETAILED DESCRIPTION:
Over the past decade, a technique widely used by ophthalmologists to assess retinal blood flow, near-infrared ICG angiography, has been applied to neurosurgical patients undergoing a wide variety of cerebrovascular procedures. This technique offers the advantage of real-time visualization of cerebral blood flow through the operating microscope at the time the procedure is being performed. Indocyanine green is an ideal agent for imaging vessels as it is tightly bound to plasma albumin, has a short half-life, and maintains an acceptable safety profile. Furthermore, the excitation and emission profiles for ICG lie in the near-infrared wavelengths, which allow penetration and imaging of vessels below a few millimeters of tissue.

Patients with either an aneurysm, compressive syndromes or pituitary and intracranial tumor will be enrolled in the study. By taking advantage of the natural fluorescence of indocyanine green (ICG) within the red spectrum and applying a light filter to the endoscope eyepiece and camera it will show as to whether this technique provides adequate visual information to differentiate perfusion in tumor and surrounding structures and to evaluate normal vessels for aneurysm and compressive syndromes procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient population would include those patients with pituitary tumors, intracranial tumors, aneurysms, and normal tissue adjacent to tumors to clarify normal from abnormal. Also, patients with compressive syndromes to ensure patency of normal vessels. This would be all patients undergoing endoscopic surgery, both endonasal and open (retromastoid or transcranial).

Exclusion Criteria:

* Less than 18 years of age
* Iodine allergy
* Shellfish allergy
* Contrast allergy
* Previous anaphylactic reaction to ICG
* Pregnant
* Anyone with any evidence of renal or hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population would include those patients with pituitary tumors, intracranial tumors, aneurysms, and normal tissue adjacent to tumors to clarify normal from abnormal. Also, patients with compressive syndromes to ensure patency of normal vessels. This would be all patients undergoing endoscopic surgery, both endonasal and open (retromastoid or transcranial).
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2015-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by observation | up to 52 weeks
  compare efficacy of tissue perfusion with and without ICG Dye and light filter

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gardner, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States